CLINICAL TRIAL: NCT01669577
Title: Independent Predictors of Mortality in Polytrauma Patients: a Prospective, Observational, Longitudinal Study
Brief Title: Independent Predictors of Mortality in Polytrauma Patients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luiz Guilherme Villares da Costa, Anesthesia division clinical staff physician, University of Sao Paulo
Other Study IDs: 1081/09
Record Dates: First submitted 2012-08-08; First posted 2012-08-21 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Trauma
Keywords: predictors; trauma; mortality
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- severe trauma patients: analysis of blood samples and clinical features
  Interventions: Procedure: analysis of blood samples and clinical features

INTERVENTIONS:
Procedure: analysis of blood samples and clinical features — clinical follow up and biochemical analysis blood at 4 time points:1-prehospital; 2-emergency room; 3- surgical center; 4-intensive care unit . 30 days follow up

SUMMARY:
Prospective observational trial searching for independent predictors of mortality. Data was collected at trauma scene, ER, three and 24 hours of hospital stay.The patients will be followed for 30 days after hospital admission.

DETAILED DESCRIPTION:
The study protocol was approved by the Institutional Medical Ethics Committee (CAPPesq 1081/09) and received financial support from the São Paulo State Research Foundation (Fundação de Amparo à Pesquisa do Estado de São Paulo - FAPESP) under no. 2010/03315-4.

At the end of data prospecting, 334 patients with severe trauma (Injury Severity Score, ISS, >15), assisted by the rescue system and taken to HCFMUSP-Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo- (by land and helicopter) were included in the study. This screening strategy included trauma patients with severe confirmed bleeding, patients with severe traumatic brain injury (TBI) and patients facing high-energy trauma (a marked characteristic of this trauma center). Patients under 18 years of age were excluded ( Figure 1).

In total, 78 patients were excluded because they did not fit the above criteria, leaving 256 patients for analysis. Of this total, 34 patients died before arriving at the emergency room, and 22 were removed from the analysis due to incomplete data, not signing the informed consent form or due to any situation in which the data collection could compromise victim care(care Figure(Figure 1).

All patients had data recorded at the following times: 1, at the trauma scene; 2, in the emergency room; 3, at 3 hours after hospital admission; and 4, at 24 hours after hospitalization.

Data regarding gender, age, trauma and trauma mechanism, medical procedures performed at all stages, time until arrival at the hospital and comorbidities were recorded. The clinical data collected were as follows: systolic blood pressure (SBP); diastolic blood pressure (DBP); heart rate (HR); respiratory rate (RR); arterial hemoglobin oxygen saturation (SAT); Glasgow Coma Scale (GCS) score; and pupil pattern. The following laboratory data were collected through peripheral venipuncture at the hospital stages: pH(hydrogenic potential); base excess (BE); bicarbonate (BIC); partial oxygen pressure (pO2); partial carbon dioxide pressure (pCO2); arterial hemoglobin oxygen saturation; lactate; sodium (Na+); potassium (K+); ionized calcium (Ca2+); glucose; hemoglobin (Hb); hematocrit (Ht); serum creatine phosphokinase (CPK); platelets and leukocytes. Data regarding volume expansion [crystalloids (CRYSTAL), colloids (COLO)], diuresis and water balance were also collected. The use of blood products [packed red blood cells (PRBC), fresh frozen plasma (FFP), platelet concentrates (PLAT), cryoprecipitate concentrates (concentrates (CRYO)] was computed, and the use of vasoactive drugs (VAD) was scored at the respective times. Patient follow-up was conducted at the intensive care unit (ICU), and time of ICU stay (days in the ICU), days under mechanic ventilation (days under MV), the presence or absence of sepsis, coagulopathy and acute renal failure (ARF) were recorded.

Blood coagulation data were collected as follows: time point 1, International Normalized Ratio (INR) and prothrombin time (PT); and time points 2, 3 and 4, INR, PT, activated partial thromboplastin time (aPTT), the respective ratio between aPTT of patients and controls (R) and thrombin time (TT).

The following severity indexes were calculated: ISS, revised trauma score (RTS); trauma and injury severity score (TRISS); and simplified acute physiology score (SAPS) 3 (the latter when the patient was in the ICU).

At time point 1, blood tests were performed using the i-STAT® device (Abbott, USA; PT/INR and CG4+ and CG8+ kits). At the hospital stages, the analyses used the clinical analysis methodology of the HCFMUSP.

Clinical follow-up was conducted for 30 days after initial trauma.

Statistical analyses The sample power analysis was conducted with a significance level of 0.05, power of 0.80, moderate correlation of 0.5 between time periods and assumption that the variability is equal within each factor (non-sphericity). Due to the effect size between 0.1 and 0.5, there was no need for samples larger than 140 patients. A total of 200 patients waswere defined conservatively, with a margin for possible deaths. The software G*Power 3.1.7 was used for sample size calculation.

The data analysis was divided into three interconnected parts. The first part refers to the descriptive data analysis and tests of association with death. The second part addressed the profiles of the time-dependent measures and their relationship with death through analysis of nonparametric variance for repeated measures. The third part includes the set of all previous analyses that resulted in a Generalized Estimating Equation (GEE).

For the first part, the analyses were performed with the overall sample (n=200) subdivided into two groups: deaths (n=52) and non-deaths (n=148). For qualitative variables, the two-tailed Fisher's exact test was used, and for quantitative variables, the two-tailed t test or the two-tailed Mann-Whitney test was used according to the normality of the variable, which was verified by the Anderson-Darling test.

In the second part, the profiles of each measure over time were analyzed for groups of survivors and non-survivors. Nonparametric analyses of variance (NPar ANOVA) were conducted.

Finally, in the third part, a GEE model was developed considering the family of binomial distributions (dichotomous response variable) with logit link function. Only the main effects of each measure were considered. The NPar ANOVA (p>0.1) was the test used for inclusion in the model. The variables for the final models were selected using the backward method, with output alpha equal to 0.05. All part 3 results were interpreted by estimating odds ratios (OR), their corresponding 95% confidence intervals and significance tests (p-value).

The significance level was set at 0.05, and the free software R 3.0.2 was used for performing the statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* severe trauma (ISS - Injury Severity Score- >15)

Exclusion Criteria:

* under 18 years old patient,
* technical problems during rescue maneuvers,
* impossibility of blood sample draw during rescue
* informed consent not provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe trauma patients evaluated at trauma scene
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luiz G Costa, MD, Principal Investigator — Hospital das Clínicas da Universidade de São Paulo
Locations (1):
- Instituto Central do Hospital das Clínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Costa LGV, Carmona MJC, Malbouisson LM, Rizoli S, Rocha-Filho JA, Cardoso RG, Auler-Junior JOC. Independent early predictors of mortality in polytrauma patients: a prospective, observational, longitudinal study. Clinics (Sao Paulo). 2017 Aug;72(8):461-468. doi: 10.6061/clinics/2017(08)02. PMID 28954004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 334 patients were collected during São Paulo rescue system activities. Entry criteria was defined as hypotensive patients (SBP<90mmHg at the scene, high-energy traumas, severe TBI); patients under 18 years old were excluded.
  If calculated ISS < 16 or no informed consent, patients were excluded.
Pre-assignment Details: Pre assignment were not performed, as patients were not known.
Groups:
- Severe Trauma Patients: intervention : analysis of blood samples
  analysis of blood samples (0,2 ml): analysis of blood samples (0,2 ml)
  analysis of blood samples: analysis of blood samples regarding electrolytes, blood gases, glucose, PT/INR collection of vital signs, blood chemistry; severity scores and intensive care unit(ICU) LOS(length of stay) were recorded
Period: Overall Study
Arm/Group | Severe Trauma Patients
Started | 334 (calculated ISS<16, no informed consent, not enough data(complete case analysis), were excluded)
Completed | 200 (complete case analysis (data missing completely at random))
Not Completed | 134
Not completed — Death | 22
Not completed — Lost to Follow-up | 78
Not completed — Physician Decision | 34

BASELINE CHARACTERISTICS:
Population: severe polytrauma patients
Groups:
- Severe Trauma Patients: Hypotensive Patients (SBP<90mmHg), severe TBI, high energy traumas All patients must have calculated ISS >15 to be included and a written informed consent should be available
Arm/Group | Severe Trauma Patients
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years]
  Continuous | 37 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 164
Region of Enrollment [Number; unit: participants]
  Brazil | 200

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: 30 days after trauma mortality evaluation
Time Frame: Within the first 30 days
Population: severe polytrauma patients (ISS>15)
Measure: Number; unit: participants
Groups:
- Severe Trauma Patients: intervention : analysis of blood samples; vital signs and clinical outcomes recorded
  analysis of blood samples (0,2 ml): analysis of blood samples (0,2 ml)
  analysis of blood samples: analysis of blood samples regarding electrolytes, blood gases, glucose, PT/INR
Arm/Group | Severe Trauma Patients
Number analyzed (Participants) | 200
participants | 52
Statistical Analysis 1: Comparison: Severe Trauma Patients; significance level of 0.05, power of 0.80, moderate correlation of 0.5 between time periods and assumption that the variability is equal within each factor (non-sphericity). Due to the effect size between 0.1 and 0.5, there was no need for samples larger than 140 patients. A total of 200 patients was defined conservatively, with a margin for possible deaths. The software G*Power 3.1.7 was used for sample size calculation. Fischer's test, Mann-Whitney, t-test; Non parametric ANOVA and GEE; Test type: Superiority or Other; p < 0.001, ANOVA — arterial hemoglobin Oxygen saturation; Non parametric(NPar) ANOVA; GEE(Generalyzed Estimation Equation) = 0.989214, 95% CI 2-sided [0.982855 to 0.995613] — GEE model (dichotomous response variable)with logit link function. The NPar ANOVA (p<0.1 for death) was the test used for inclusion in the model variables for the final models - backward method, with alpha equal to 0.05
Statistical Analysis 2: Comparison: Severe Trauma Patients; diastolic arterial blood pressure; Test type: Superiority or Other; p < 0.001, ANOVA; GEE = 0.997280, 95% CI 2-sided [0.995791 to 0.998772]
Statistical Analysis 3: Comparison: Severe Trauma Patients; lactate; Test type: Superiority or Other; p < 0.004, ANOVA; GEE = 1.046961, 95% CI 2-sided [1.012521 to 1.082572]
Statistical Analysis 4: Comparison: Severe Trauma Patients; Glasgow coma score; Test type: Superiority or Other; p < 0.001, ANOVA; GEE = 0.973987, 95% CI 2-sided [0.965308 to 0.982744]
Statistical Analysis 5: Comparison: Severe Trauma Patients; amount of Infused crystalloids; Test type: Superiority or Other; p < 0.023, ANOVA; GEE = 1.000013, 95% CI 2-sided [1.000000 to 1.000025]

ADVERSE EVENTS:
Time Frame: 30 days follow up
Description: Patients were monitored for adverse outcomes related to venipuncture, as this was the unique intervention.
Groups:
- Severe Trauma Patients: intervention : analysis of blood samples
  analysis of blood samples (0,2 ml): analysis of blood samples (0,2 ml)
  analysis of blood samples: analysis of blood samples regarding electrolytes, blood gases, glucose, PT/INR
Arm/Group | Severe Trauma Patients
Serious Adverse Events (participants affected / at risk) | 1/200
Other Adverse Events (participants affected / at risk) | 2/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Trauma Patients (N=200)
Thrombophlebitis (Vascular disorders) | 1 (1) — 1 patient was diagnosed by ultrasound and persistent positive blood cultures. Another foci of infection were discarded and patient treated with antibiotics and systemic anticoagulation( iv non fractionated heparin) until resolution of septic state.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Trauma Patients (N=200)
Infection (Infections and infestations) | 2 (2) — 2 patients had skin infection at the peripheral venous acess site (performed at the prehospital stage)

LIMITATIONS AND CAVEATS:
single center trial, majority of TBI and male patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No